CLINICAL TRIAL: NCT04041284
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Followed by an Open-Label Extension to Evaluate the Efficacy and Safety of Fremanezumab for Preventive Treatment of Migraine in Patients With Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Fremanezumab for Preventive Treatment of Migraine in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TV48125-MH-40142; 2019-001989-15 (EudraCT Number)
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Migraine; Major Depressive Disorder
MeSH Terms: conditions — Migraine Disorders; Depressive Disorder, Major | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- fremanezumab (Experimental): monthly 225 mg. In the open-label extension phase starting at week 12, all participants will receive active treatment with a quarterly dose of 675 mg sc
  Interventions: Drug: Fremanezumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Monthly 225 mg subcutaneous
  Other Names: TEV-48125, LBR-101, PF-04427429, RN307
  Arms: fremanezumab
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy of monthly 225 mg sc fremanezumab in adult participants with migraine and major depressive disorder (MDD)

The secondary objectives are to evaluate the efficacy of monthly 225 mg sc of fremanezumab in adult participants with migraine and MDD on the reduction of MDD symptoms, responder rates in monthly migraine days, improving quality of life, improving disability, and the safety and tolerability of monthly 225 mg sc and quarterly 675 mg sc fremanezumab in adult participants with migraine and MDD.

The total duration of participant participation in the study is planned to be approximately 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine with onset at ≤50 years of age.
* Prior to the screening visit 1 the participant has a 12-month history of either migraine or headache consistent with migraine
* The participant agrees not to initiate any migraine preventive during the study. Up to 30% of participants, however, may take a single such medication previously prescribed for the treatment of migraine.
* The participant has a history of major depressive disorder (MDD) at least 12 months prior to the screening visit. Participants may take a single medication prescribed for the treatment of depression as long as the dose of that medication has been stable for at least 8 weeks prior to the screening visit and expects to remain at the stable dose throughout the study.
* The participant has a body weight ≥ 45 kg and a body mass index within the range of 17.5 to 34.9 kg/m2, inclusive.
* Women of child-bearing potential whose male partners are potentially fertile (ie, no vasectomy) must use highly effective birth control methods for the duration of the study and for 6 months after discontinuation of IMP.
* Men must be sterile or, if they are potentially fertile/reproductively competent (not congenitally sterile) and their female partners are of child-bearing potential, must use a condom for the duration of the study and for 6 months after discontinuation of IMP.

NOTE: Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has failed 4 or more different medication classes to treat depression in their lifetime.
* The participant has used an intervention/device (eg, scheduled nerve blocks, implantable vagal nerve stimulation, and transcranial magnetic stimulation) for migraine or depression during the 2 months prior to screening.
* The participant has used electroconvulsive therapy at any time.
* The participant suffers from constant or nearly constant headache, defined as having headaches for more than 80% of the time he/she is awake, and less than 4 days without headache per month. Daily headache is acceptable if participant has headaches 80% or less of the time he/she is awake on most days.
* The participant has a clinical history of a severe or uncontrolled psychiatric disorder, to include the following, or at the discretion of the investigator for any clinically significant psychiatric history that would likely interfere with full participation in the study:

  * Lifetime exclusion: suicide attempt
  * In the past 6 months exclusion: suicidal ideation, or other psychoactive spectrum disorders including schizoaffective disorder, delusional disorder, depression with psychotic features, and catatonic disorder.
* The participant has a known infection or history of human immunodeficiency virus, tuberculosis, any history of Lyme disease, or chronic hepatitis B or C infection.
* The participant has a past or current history of cancer, except for appropriately treated non-melanoma skin carcinoma.
* The participant is a pregnant or nursing female or plans to become pregnant during the study, including the 6-month period after the administration of the last dose.
* The participant has a history of hypersensitivity reactions to injected proteins, including monoclonal antibodies, or a history of Stevens-Johnson Syndrome or toxic epidermal necrolysis syndrome.
* Participant has received onabotulinumtoxinA for migraine or for any medical or cosmetic reasons requiring injections in the head, face, or neck during the 3 months before screening visit.
* The participant has a history of hypersensitivity reactions to injected proteins, including monoclonal antibodies.
* The participant has participated in a clinical study of a new chemical entity or a prescription medicine within 2 months of the screening visit or 3 months in case of biologics if the half-life of the biologics is unknown or 5 half-lives, whichever is longer, or is currently participating in another study of an IMP (or a medical device).
* The participant has failed treatment (based on tolerability and/or a lack of efficacy) with any monoclonal antibodies targeting the CGRP pathway (erenumab, eptinezumab, galcanezumab, or fremanezumab) or have taken the medications within 5 half-lives of the screening visit (V1) or take them during the study.
* The participant has any clinically significant uncontrolled medical condition (treated or untreated).
* The participant has a history of alcohol or drug abuse in the opinion of the investigator.
* The participant has evidence or medical history of psychotic symptoms as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria such as delusions, hallucinations, or disorganized speech in the past 1 month.

NOTE: Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (64):
- United States (17):
  - Teva Investigational Site 14330, Little Rock, Arkansas
  - Teva Investigational Site 14337, San Diego, California
  - Teva Investigational Site 14342, Denver, Colorado
  - Teva Investigational Site 14332, Stamford, Connecticut
  - Teva Investigational Site 14329, Hialeah, Florida
  - Teva Investigational Site 14334, Jacksonville, Florida
  - Teva Investigational Site 14341, Orlando, Florida
  - Teva Investigational Site 14411, Tampa, Florida
  - Teva Investigational Site 14336, Pikesville, Maryland
  - Teva Investigational Site 14331, Waltham, Massachusetts
  - Teva Investigational Site 14343, Bolivar, Missouri
  - Teva Investigational Site 14335, Brooklyn, New York
  - Teva Investigational Site 14345, The Bronx, New York
  - Teva Investigational Site 14340, Portland, Oregon
  - Teva Investigational Site 14338, Philadelphia, Pennsylvania
  - Teva Investigational Site 14333, Memphis, Tennessee
  - Teva Investigational Site 14339, Nashville, Tennessee
- Czechia (5):
  - Teva Investigational Site 54190, Choceň
  - Teva Investigational Site 54183, Prague
  - Teva Investigational Site 54184, Prague
  - Teva Investigational Site 54185, Prague
  - Teva Investigational Site 54186, Rychnov nad Kněžnou
- Finland (4):
  - Teva Investigational Site 40058, Kuopio
  - Teva Investigational Site 40057, Oulu
  - Teva Investigational Site 40056, Tampere
  - Teva Investigational Site 40055, Turku
- France (2):
  - Teva Investigational Site 35265, Bron
  - Teva Investigational Site 35267, Saint-Priest-en-Jarez
- Germany (6):
  - Teva Investigational Site 32736, Dresden
  - Teva Investigational Site 32737, Essen
  - Teva Investigational Site 32731, Essen
  - Teva Investigational Site 32734, Leipzig
  - Teva Investigational Site 32732, Mittweida
  - Teva Investigational Site 32733, Westerstede
- Greece (3):
  - Teva Investigational Site 63075, Athens
  - Teva Investigational Site 63076, Glyfada
  - Teva Investigational Site 63077, Marousi
- Israel (5):
  - Teva Investigational Site 80172, Hadera
  - Teva Investigational Site 80173, Holon
  - Teva Investigational Site 80177, Jerusalem
  - Teva Investigational Site 80178, Petah Tikva
  - Teva Investigational Site 80175, Rehovot
- Italy (6):
  - Teva Investigational Site 30242, Catanzaro
  - Teva Investigational Site 30236, Florence
  - Teva Investigational Site 30237, Milan
  - Teva Investigational Site 30235, Pavia
  - Teva Investigational Site 30232, Roma
  - Teva Investigational Site 30234, Rome
- Poland (4):
  - Teva Investigational Site 53447, Krakow
  - Teva Investigational Site 53445, Poznan
  - Teva Investigational Site 53446, Warsaw
  - Teva Investigational Site 53448, Wroclaw
- Russia (4):
  - Teva Investigational Site 50482, Moscow
  - Teva Investigational Site 50483, Moscow
  - Teva Investigational Site 50480, Moscow
  - Teva Investigational Site 50481, Nizhny Novgorod
- Spain (4):
  - Teva Investigational Site 31276, Seville
  - Teva Investigational Site 31274, Valencia
  - Teva Investigational Site 31272, Valladolid
  - Teva Investigational Site 31273, Zaragoza
- Ukraine (3):
  - Teva Investigational Site 58319, Kiyv
  - Teva Investigational Site 58321, Odesa
  - Teva Investigational Site 58320, Vinnytsia
- Teva Investigational Site 34254, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Lipton RB, Ramirez Campos V, Roth-Ben Arie Z, Galic M, Mitsikostas D, Tassorelli C, Denysenko L, Cohen JM. Fremanezumab for the Treatment of Patients With Migraine and Comorbid Major Depressive Disorder: The UNITE Randomized Clinical Trial. JAMA Neurol. 2025 Jun 1;82(6):560-569. doi: 10.1001/jamaneurol.2025.0806. PMID 40323613

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 540 participants screened, 353 participants were enrolled/randomized.
Groups:
- Placebo: Participants received placebo matched to fremanezumab subcutaneously (SC) during the 12-week double blind (DB) period and then continued into the open-label (OL) extension period in which all participants received a single quarterly dose of fremanezumab Dose 2 SC on Day 85.
- Fremanezumab: Participants received monthly doses of fremanezumab Dose 1 SC during the 12-week DB period and then continued into the OL extension period in which all participants received a single quarterly dose of fremanezumab Dose 2 SC on Day 85.
Period: DB Phase (12 Weeks)
Arm/Group | Placebo | Fremanezumab
Started | 178 | 175
DB Safety Analysis Set (All randomized participants who received at least 1 dose of study drug during the DB treatment period.) | 177 | 176 (One participant was randomized to Placebo and received placebo in the DB period but was summarized in the Fremanezumab treatment group in all safety summaries due to an error in recording treatment.)
DB Modified Intent-to-treat (mITT) Analysis Set (All randomized participants who received at least 1 dose of study drug and had at least 10 days of postrandomization efficacy assessment on the primary endpoint.) | 178 | 175
Completed | 166 | 164
Not Completed | 12 | 11
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Protocol deviation | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other than specified | 1 | 0
Period: OL Phase (12 Weeks)
Arm/Group | Placebo | Fremanezumab
Started | 166 | 164
OL Safety Analysis Set (All participants who received at least 1 of dose of study drug during the OL treatment period.) | 165 | 165 (One participant was randomized to Placebo and received placebo in the DB period but was summarized in the Fremanezumab treatment group in all safety summaries due to an error in recording treatment.)
OL mITT Analysis Set (All participants who received at least 1 dose of study drug during the OL treatment period and had at least 10 days of diary entries during the OL period.) | 165 | 161
Completed | 154 | 155
Not Completed | 12 | 9
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Protocol deviation | 0 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Other than specified | 6 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: Participants received placebo matched to fremanezumab SC during the 12-week DB period and then continued into the OL extension period in which all participants received a single quarterly dose of fremanezumab Dose 2 SC on Day 85.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab | Total
Number analyzed (Participants) | 178 | 175 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.64) | 43.5 (11.94) | 42.9 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 154 | 310
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 171 | 170 | 341
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 172 | 170 | 342
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Number of migraine days [Mean (Standard Deviation); unit: days] — A migraine day was defined as when at least 1 of following occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine (where only 1 migraine criterion was missing); demonstrating a headache of any duration that was treated with migraine-specific medications; and a calendar day that was immediately consecutive of any day fulfilling the 3 criteria above, where participants report headache of any duration.
  days | 14.4 (6.15) | 15.1 (6.41) | 14.8 (6.28)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Average Number of Migraine Days During the 12-Week DB Treatment Phase After the First Dose of Study Drug
Description: A migraine day was defined as when at least 1 of following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine (where only 1 migraine criterion was missing); a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds); and a calendar day (00:00 to 23:59) that was immediately consecutive of any day fulfilling 3 criteria above, where participants report headache of any duration. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12 week period/number of days with assessments recorded in e-diary for 12 week period)*28. Least square (LS) mean was calculated using analysis of covariance (ANCOVA).
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: DB mITT analysis set included all randomized participants who received at least 1 dose of study drug and had at least 10 days of postrandomization efficacy assessment on the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: days
Groups:
- Double-blind Phase: Placebo: Participants received placebo matched to fremanezumab SC during the 12-week DB period.
- Double-blind Phase: Fremanezumab: Participants received monthly doses of fremanezumab Dose 1 SC during the 12-week DB period.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
days | -2.9 (0.49) | -5.1 (0.50)
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p < 0.0001, ANCOVA; LS mean difference = -2.2, 95% CI 2-sided [-3.16 to -1.21], Standard Error of Mean 0.50

2. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale-17 (HAM-D 17) Items Total Score at Week 8
Description: The HAM-D 17 is a list of 17 items used to determine a participant's level of depression. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 (none/absent) to 2 (severe symptom) include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 (none/absent) to 4 (severe symptom): Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The HAM-D17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAM-D17 scores indicate more severe depression. LS mean was calculated using mixed-effects model for repeated measures (MMRM).
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
units on a scale | -4.6 (0.54) | -6.0 (0.55)
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p = 0.0205, Mixed Models Analysis; LS mean difference = -1.4, 95% CI 2-sided [-2.61 to -0.22], Standard Error of Mean 0.61

3. Secondary Outcome: Number of Participants With ≥50% Reduction in Monthly Average Number of Migraine Days During the 12 Weeks After the First Dose of Study Drug
Description: A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds); and a calendar day (00:00 to 23:59) that was immediately consecutive of any day fulfilling the 3 criteria above, where participants report headache of any duration. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12 week period/number of days with assessments recorded in e-diary for 12 week period)*28.
Time Frame: Baseline (Day -28 to Day -1) up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
Participants | 24 | 57
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.89 to 5.62]

4. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life (MSQoL) Questionnaire Role Function-Restrictive and Role Function-Preventive Domain Scores at Week 12
Description: The MSQoL version 2.1 is a 14-item questionnaire that assesses the impact of migraine and migraine treatment on a participant's quality of life during the previous 4 weeks. Each item is scored on a 6-point scale where: 1=none of the time to 6=all of the time. The MSQoL measures the degree to which performance of normal activities is limited by migraine (Role Function-Restrictive domain comprising 7 items; score range 7 to 42), the degree to which performance of normal activities is prevented by migraine (Role Function-Preventive domain comprising 4 items; score range 4 to 24), and the emotional effects of migraine (Emotional Function domain comprising 3 items; score range 3 to 18). Total raw scores for each domain is the sum of the final item value for all of the items in that domain. After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health-related quality of life. LS mean was calculated using MMRM.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
units on a scale
  Restrictive score | 15.9 (2.00) | 27.2 (2.04)
  Preventive score | 12.3 (1.95) | 22.2 (2.00)
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p < 0.0001, Mixed Models Analysis; LS mean difference = 11.3, 95% CI 2-sided [6.91 to 15.59], Standard Error of Mean 2.21 — Restrictive score: Fremanezumab versus placebo
Statistical Analysis 2: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p < 0.0001, Mixed Models Analysis; LS mean difference = 9.9, 95% CI 2-sided [5.73 to 14.08], Standard Error of Mean 2.12 — Preventive score: Fremanezumab versus placebo

5. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Scale Score at Weeks 4, 8, and 12
Description: The CGI-S is a short questionnaire filled out by the investigator that rates a participant's mental health from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
units on a scale
  Change at Week 4 | -0.4 (0.10) | -0.6 (0.10)
  Change at Week 8 | -0.6 (0.10) | -0.1 (0.10)
  Change at Week 12 | -0.8 (0.10) | -1.1 (0.10)
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p = 0.0915, Mixed Models Analysis; LS mean difference = -0.2, 95% CI 2-sided [-0.39 to 0.03], Standard Error of Mean 0.11 — Change at Week 4: Fremanezumab versus Placebo
Statistical Analysis 2: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p = 0.0006, Mixed Models Analysis; LS mean difference = -0.4, 95% CI 2-sided [-0.59 to -0.16], Standard Error of Mean 0.11 — Change at Week 8: Fremanezumab versus Placebo
Statistical Analysis 3: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p = 0.0030, Mixed Models Analysis; LS mean difference = -0.4, 95% CI 2-sided [-0.58 to -0.12], Standard Error of Mean 0.12 — Change at Week 12: Fremanezumab versus Placebo

6. Secondary Outcome: Change From Baseline in 6-Item Headache Impact Test (HIT-6) Disability Score at Week 12
Description: Migraine related disability was assessed using the HIT-6. The questionnaire measures the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning, and psychological distress. It also assesses headache severity. Each question was answered on the scale ranging with the following response options: 6 points (never), 8 points (rarely), 10 points (sometimes), 11 points (very often), and 13 points (always). The total score was obtained from summation of the 6 question points. The HIT-6 total score ranges between 36 and 78, with higher scores reflecting greater impact.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab
Number analyzed (Participants) | 178 | 175
units on a scale | -5.2 (0.71) | -8.8 (0.73)
Statistical Analysis 1: Comparison: Double-blind Phase: Placebo vs Double-blind Phase: Fremanezumab; Test type: Other; p < 0.0001, Mixed Models Analysis; LS mean difference = -3.6, 95% CI 2-sided [-5.15 to -1.96], Standard Error of Mean 0.81

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered TEAEs if onset occurred on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 24
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period.
  OL safety analysis set included all participants who received at least 1 of dose of study drug during the OL treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Phase: Placebo/Fremanezumab Dose 2; Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2: Participants received a single quarterly dose of fremanezumab Dose 2 SC on Day 85.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants | 48 | 70 | 31 | 29

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Criteria for potentially clinically significant vital signs values: Pulse: ≥120 beats per minute (bpm) and increase from baseline of ≥15 bpm or ≤50 bpm and decrease from baseline of ≥15 bpm; Systolic blood pressure (SBP): ≥180 millimeters of mercury (mmHg) and increase from baseline of ≥20 mmHg or ≤90 mmHg and decrease from baseline of ≥20 mmHg; Diastolic blood pressure (DBP): ≥105 mmHg and increase from baseline of ≥15 mmHg or ≤50 mmHg and decrease from baseline of ≥15 mmHg; Respiratory rate: <10 breaths per minute; and Body temperature: ≥38.3 degrees celsius (ºC) and change from baseline of ≥1.1ºC.
Time Frame: Baseline up to Week 24
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period.
  OL safety analysis set included all participants who received at least 1 of dose of study drug during the OL treatment period.
  Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 174 | 173 | 162 | 164
Participants | 0 | 5 | 2 | 1

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Physical Examination Findings
Description: Physical examination included height, weight, general appearance; head, eyes, ears, nose, and throat; chest and lungs; heart; abdomen; musculoskeletal; skin; lymph nodes; and neurological. Clinical significance was per investigator's discretion.
Time Frame: Baseline up to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Drug Hypersensitivity and Seasonal Allergy
Time Frame: Baseline up to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants
  Drug hypersensitivity | 0 | 1 | 0 | 0
  Seasonal allergy | 1 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants Who Used Concomitant Medication
Description: Concomitant medications included agents acting on the renin-angiotensin system, analgesics, antibacterials for systemic use, antihistamines for systemic use, anti-inflammatory and antirheumatic products, beta-blocking agents, drugs for acid related disorder, lipid modifying agents, mineral supplement, other gynecologicals, psychoanaleptics, psycholeptics, sex hormones and modulators of the genital system, thyroid therapy, vaccines, and vitamins.
Time Frame: Baseline up to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants | 173 | 173 | 160 | 163

12. Secondary Outcome: Number of Participants Who Used Concomitant Medication for Migraine/Headache
Description: Concomitant medications for migraine/headache included analgesics, antiepileptics, muscle relaxants, anti-inflammatory and antirheumatic products, agents acting on the renin-angiotensin system, anesthetics, antianemic preparations, antibacterials for systemic use, antihistamines for systemic use, beta-blocking agents, lipid modifying agents, mineral supplement, other gynecologicals, psychoanaleptics, psycholeptics, sex hormones and modulators of the genital system, thyroid therapy, vaccines, vitamins etc.
Time Frame: Baseline up to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants | 170 | 169 | 156 | 160

13. Secondary Outcome: Number of Participants Who Did Not Complete the Study Due to AE
Time Frame: Baseline up to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 165 | 165
Participants | 0 | 3 | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Any Suicidal Ideation or Suicidal Behavior According to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS included responses for Suicidal Ideation or Suicidal Behavior in 10 categories: 1=Wish to be dead; 2=Non-specific active suicidal thoughts; 3=Active suicidal ideation with any methods (not plan) without intent to act; 4=Active suicidal ideation with some intent to act, without specific plan; 5=Active suicidal ideation with specific plan and intent; 6=Preparatory acts or behavior; 7=Aborted attempt; 8=Interrupted attempt; 9=Non-fatal suicide attempt; and 10=Completed suicide. Participants who responded "Yes" to any category were considered Positive, participants who responded "No" for all categories were considered Negative, and participants who were evaluable but did not complete the questionnaire were considered Incomplete. A Positive response was considered as a worse outcome and the investigator determined if further evaluation was needed. Any Suicidal ideation or Suicidal Behavior events reported as TEAEs along with all other reported TEAEs are included in the AE module.
Time Frame: Baseline, Weeks 4, 8, 12, and 24
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint of the respective phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
Number analyzed (Participants) | 177 | 176 | 153 | 155
Participants
  Baseline: number analyzed (Participants) | 177 | 176 | 0 | 0
  Baseline: Incomplete | 0 | 0 |  |
  Baseline: Negative | 177 | 176 |  |
  Baseline: Positive | 0 | 0 |  |
  Week 4: number analyzed (Participants) | 169 | 169 | 0 | 0
  Week 4: Incomplete | 1 | 0 |  |
  Week 4: Negative | 168 | 168 |  |
  Week 4: Positive | 0 | 1 |  |
  Week 8: number analyzed (Participants) | 170 | 164 | 0 | 0
  Week 8: Incomplete | 0 | 0 |  |
  Week 8: Negative | 170 | 164 |  |
  Week 8: Positive | 0 | 0 |  |
  Week 12: number analyzed (Participants) | 165 | 163 | 0 | 0
  Week 12: Incomplete | 0 | 0 |  |
  Week 12: Negative | 165 | 163 |  |
  Week 12: Positive | 0 | 0 |  |
  Week 24: number analyzed (Participants) | 0 | 0 | 153 | 155
  Week 24: Incomplete |  |  | 0 | 0
  Week 24: Negative |  |  | 152 | 153
  Week 24: Positive |  |  | 1 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period. OL safety analysis set included all participants who received at least 1 of dose of study drug during the OL treatment period.
  One participant was randomized to Placebo and received placebo in the DB period but was summarized in the Fremanezumab treatment group in all safety summaries due to an error in recording treatment.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Fremanezumab | Open-label Phase: Placebo/Fremanezumab Dose 2 | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/176 | 0/165 | 0/165
Serious Adverse Events (participants affected / at risk) | 1/177 | 2/176 | 3/165 | 1/165
Other Adverse Events (participants affected / at risk) | 0/177 | 0/176 | 0/165 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Phase: Placebo (N=177) | Double-blind Phase: Fremanezumab (N=176) | Open-label Phase: Placebo/Fremanezumab Dose 2 (N=165) | Open-label Phase: Fremanezumab Dose 1/Fremanezumab Dose 2 (N=165)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT04041284/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04041284/SAP_001.pdf